CLINICAL TRIAL: NCT04159181
Title: Investigations of the Endocrine Colon in Healthy Individuals
Brief Title: The Endocrine Colon in Humans
Acronym: Colon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Simon Veedfald, Investigator, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CBC-COLON-18
Record Dates: First submitted 2018-07-09; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: Colon; PYYs; GLP-1; Gut peptides; Fermentation; Lactulose; human
MeSH Terms: interventions — Lactulose; picosulfate sodium; Water

STUDY DESIGN:
Intervention Model Description: Healthy men studied on three occasions. Study A and B will be conducted in random order. Day C wil always be conducted as the last study day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Day A (Experimental): After an overnight fast participants will receive an oral solution of lactulose (20g lactulose/200mL water).
  Interventions: Other: Lactulose
- Day B (Experimental): After an overnight fast participants will drink 200mL of water
  Interventions: Other: Placebo (water)
- Day C (Experimental): After an overnight fast and an evacuation of the colonic content, participants will receive an oral solution of lactulose (20g lactulose/200mL water).
  Interventions: Other: Lactulose; Other: Picoprep

INTERVENTIONS:
Other: Lactulose — Oral solution lactulose (20g lactulose/200mL water).
  Arms: Day A; Day C
Other: Picoprep — Cathartic to accomplish an evacuation of the colonic content.
  Arms: Day C
Other: Placebo (water) — oral administration of Water (200mL).
  Arms: Day B

SUMMARY:
This study will examine the role of the colon as an endocrine organ with a focus on the secretion of gastrointestinal peptides.

DETAILED DESCRIPTION:
This study will examine the role of the colon as an endocrine organ with a focus on the secretion of gastrointestinal peptides.

We aim to determine the contribution of the colon to the fasting and postprandial release of gut peptides such as glucagon-like peptide-1 (GLP-1) and peptide YY (PYY). Young healthy men will be examined on three occasions at a clinical research Facility after an overnight fast. On one occasion the colon will also be emptied using a cathartic (picoprep). On two occasions an oral solution of lactulose will be administered to stimulate fermentation by colonic bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young men (self-reported)
* BMI between 18,5-24,9 kg/m^2

Exclusion Criteria:

* Diabetes mellitus (elevated fasting plasma glucose or HbA1c)
* Family history of diabetes mellitus
* Intestinal disease (e.g. inflammatory bowel disease, malabsorption)
* Family history of intestinal diseases
* Previous gastrointestinal surgery
* BMI >25 kg/m^2
* Tobacco use
* Alcohol consumption > 14 standard drinks/week
* Drug use
* Kidney, Heart- or Liver disease
* Treatment with prescription drugs that can not be held for 12h
* Constipation
* Accelerated or delayed gastric emptying
* Absence of daily bowel movements
* Vegetarian lifestyle
* > than 3kgs weightloss or weight gain within 3 months
* Haemoglobin concentration < 8,0mmol/L
* Bleeding diathesis
* Latex or bandaid allergies

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
GLP-1 | -60, -45, -30, -15, 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240, 255, 270. 285, 300 min
  Plasma concentrations of glucagon-like peptide-1 (GLP-1)

SECONDARY OUTCOMES:
PYY | -60, -45, -30, -15, 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240, 255, 270. 285, 300 min
  Plasma concentrations of peptide YY (PYY)
Hydrogen breath test | -60, -45, -30, -15, 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240, 255, 270. 285, 300 min
  Concentrations of hydrogen in exhaled air
Ghrelin | -60, -45, -30, -15, 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240, 255, 270. 285, 300 min
  Plasma concentrations of ghrelin
Motilin | -60, -45, -30, -15, 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240, 255, 270. 285, 300 min
  Plasma concentrations of motilin
Neurotensin | -60, -45, -30, -15, 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240, 255, 270. 285, 300 min
  Plasma concentrations of Neurotensin
Glucagon | -60, -45, -30, -15, 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240, 255, 270. 285, 300 min
  Plasma concentrations of glucagon

CONTACTS AND LOCATIONS:
Overall Officials: Jens J Holst, MD, Dr.med., Study Director — University of Copenhagen
Locations (2):
- Denmark (2):
  - University of Copenhagen, Copenhagen, Capital
  - Hvidovre University Hospital, Hvidovre, Capital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christiansen CB, Veedfald S, Hartmann B, Gauguin AM, Moller S, Moritz T, Madsbad S, Holst JJ. Colonic Lactulose Fermentation Has No Impact on Glucagon-like Peptide-1 and Peptide-YY Secretion in Healthy Young Men. J Clin Endocrinol Metab. 2022 Jan 1;107(1):77-87. doi: 10.1210/clinem/dgab666. PMID 34508600